CLINICAL TRIAL: NCT03534505
Title: A Prospective Randomized Controlled Double-Blind of Post-Operative Analgesic Effects of Local Wound Infiltration With Ketorolac After Inguinal Herniorrhaphy
Brief Title: Post-Operative Analgesic Effects of Local Wound Infiltration With Ketorolac After Inguinal Herniorrhaphy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: cannot enroll patient
Sponsor: Mahidol University (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/456
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Inguinal Herniorrhaphy; Pain, Postoperative
Keywords: Inguinal Herniorrhaphy; Analgesic Effects of Local Wound
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Once given general anesthesia in the operating room, the patient will be randomly selected into one of the two arms of this report's diagram (1:1 ratio) through the drawing of a sealed, opaque envelope by one of the surgical residents in charge or by the attending surgeon. All patients will undergo herniorrhaphy with Lichtenstein Tension-Free Repair technique. After abdominal sheath will be closed by Vicryl No.0, Patients who are the Ketorolac group will receive local infiltration in abdominal sheath layer with Ketorolac 30 mg in normal saline 10ml. and patients who are the control group will receive local infiltration with 0.5% bupivacaine 10 ml. And then skin closure will be done by nylon 3-0.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac injections (Experimental): Patients will undergo herniorrhaphy with Lichtenstein Tension-Free Repair technique. After abdominal sheath will be closed by Vicryl No.0, Patients who are the Ketorolac group will receive local infiltration in abdominal sheath layer with Ketorolac 30 mg in normal saline 10ml. And then skin closure will be done by nylon 3-0.
  Interventions: Other: Ketorolac group
- bupivacaine (Active Comparator): Patients will undergo herniorrhaphy with Lichtenstein Tension-Free Repair technique. After abdominal sheath will be closed by Vicryl No.0, Patients who are the bupivacaine group will receive local infiltration in abdominal sheath layer with 0.5% bupivacaine 10 ml. And then skin closure will be done by nylon 3-0.
  Interventions: Other: Bupivacaine group

INTERVENTIONS:
Other: Ketorolac group — patients will undergo herniorrhaphy with Lichtenstein Tension-Free Repair technique. After abdominal sheath will be closed by Vicryl No.0, Patients who are the Ketorolac group will receive local infiltration in abdominal sheath layer with Ketorolac 30 mg in normal saline 10ml. And then skin closure will be done by nylon 3-0.
  Arms: Ketorolac injections
Other: Bupivacaine group — patients will undergo herniorrhaphy with Lichtenstein Tension-Free Repair technique. After abdominal sheath will be closed by Vicryl No.0, Patients who are the Bupivacaine group will receive local infiltration in abdominal sheath layer with 0.5% bupivacaine 10 ml. And then skin closure will be done by nylon 3-0.
  Arms: bupivacaine

SUMMARY:
Inguinal hernia is one of the most common diseases worldwide, including Thailand. Patients who underwent treatment of inguinal hernia (herniorrhaphy) found surgical site pain.There are many procedures to relieve pain after surgery. Injection of pain killer at the surgical site is a well-known method nowadays, especially with NSAIDs; Nowadays, Ketorolac is among the most-often used drug in the research. B. Ben-David's et al. published in 1995. is the study of the effects of the Ketorolac by comparing 60 mg of Ketorolac injected intramuscularly and 30 mg injections at the surgical site in 32 patients who underwent herniorrhaphy. Observing patients after surgery, postoperative pain score at 2 and 6. After 24 hours of surgery, they found that the patients who were given Ketorolac 30 mg suffered less pain than the group of patients who had Ketorolac 60 mg with statistical significant (P<0.05). The study by Connelly and colleagues, published in 1997, was a randomized double-blind study which compared the performance of relieving pain after surgery of surgical site injection of Ketorolac 60 mg and intravenous injection of Ketorolac 60 mg. In studies of 30 patients with herniorrhaphy surgery, the results showed within 24 hours of surgery, the group of patients with surgical site injections suffered less pain than the group of patients with intravenous injection (P<0.02). Besides they discovered that the time to first analgesia in the group of patients with surgical site injection was longer. (P<0.03), and the amount of analgesic requirement that the patients needed in the first 24 hours after surgery was also less in this group. (P<0.0002). According to the research above surgical site injection of Ketorolac is effective in pain relief. Bupivacaine is the most accepted drug using local infiltratively to relieve the pain especially in patients with herniorrhaphy. Previous studies of Bupivacaine found that Bupivacaine is a very effective in pain reliever, can reduce the usage of opioids, and also can reduce the recovery time in hospital. Thus, our study is to demonstrate the effectiveness of pain relief after surgery by local infiltration of Ketorolac in a patients who undergo herniorrhaphy by dividing patients into two groups and comparing between Ketorolac and Bupivacaine injection at surgical site.

DETAILED DESCRIPTION:
The study design is a prospective randomized, double-blind, controlled trial of patients who are undergoing elective unilateral inguinal herniorrhaphy at Ramathibodi Hospital during the period 1 July 2018 - 30 June 2020 The primary outcome is to study the effectiveness of Ketorolac injections in pain relief after herniorrhaphy surgery and the secondary outcome is to study the adverse effects and complications after injection of Ketorolac: anaphylactic shock, abnormal bleeding at surgical wound, gastrointestinal bleeding and acute kidney injury.

After approval by the ethics committee, patients scheduled for elective unilateral inguinal herniorrhaphy under general anesthesia who are eligible for inclusion criteria will be recruited for this study after informed consent by surgical residents or surgical staff at the Out Patient Department (OPD). Patients who meet the exclusion criteria will be excluded.

During a preoperative visit, the patients will be introduced to the concept of the visual analogue scale (VAS), which ranges from 0 = no pain to 10 = worst pain.

Once given general anesthesia in the operating room, the patient will be randomly selected into one of the two arms of this report's diagram (1:1 ratio) through the drawing of a sealed, opaque envelope by one of the surgical residents in charge or by the attending surgeon. All patients will undergo herniorrhaphy with Lichtenstein Tension-Free Repair technique. After abdominal sheath will be closed by Vicryl No.0, Patients who are the Ketorolac group will receive local infiltration in abdominal sheath layer with Ketorolac 30 mg in normal saline 10 ml. and patients who are the control group will receive local infiltration with 0.5% bupivacaine 10 ml. And then skin closure will be done by nylon 3-0.

A standardized plan for postoperative analgesia is prepared. All patients will receive one 500 mg tablet of oral paracetamol every 6 hours when postoperative oral intake is allowed by the attending doctor. In patients with VAS scores >3, parenteral opioid (Morphine) is given.

The hospital volunteer nurses caring for the patients during the preoperative and postoperative course are given standard pain evaluation protocols. All study pain evaluators and patients are blinded to treatment assignments throughout the pain assessment process.

After the operation, the inpatient ward nurse will record the patients' pain scores at 4,8, and 12 hours after surgery using the VAS score and record the results in the study data recording form attached to each patient's medical record chart. Additional morphine usage data is also recorded.

All adverse effects and complications after injection of Ketorolac injection such as anaphylactic shock, abnormal bleeding at surgical wound, gastrointestinal bleeding and acute kidney injury will be recorded and treated by the attending resident or consultant doctor. All data is collected by the main investigator from the patient chart and data recording form. Data is expressed as mean ± SD. Parametric data is compared between groups. Statistical significance is set at a level of p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years old undergoing elective unilateral inguinal herniorrhaphy at Ramathibodi hospital
* Patients who are ASA classification 1-2
* Patients who had normal liver function test : AST 5-34 U/L , ALT 0-55 U/L, ALP 40-150 U/L ,TB0.2-1.2 mg/dL ,DB 0.0-0.5 mg/dL
* Patients who are going the operation under general anesthesia
* Patients who undergoing herniorrhaphy with Lichtenstein Tension-Free Repair technique

Exclusion Criteria:

* Patients who had femoral hernia
* Patients who had history of NSAIDs allergy
* Patients with history of prior hernorrhaphy
* Patients who had history of GI bleeding and gastritis
* Patients who had infection
* Patients who had history of SLE, HIV, asthma , cardiovascular disease and chronic kidney disease(GFR<60 ml/min/1.73m2)
* Patients with end stage disease
* Patients who are pregnant
* Patients who reject or withdrawal from research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Ketorolac injections in term of pain at 4 hours using visual analog scale after herniorrhaphy surgery. | 4 hours
  Effectiveness of Ketorolac injections in term of pain using visual analog scale after herniorrhaphy surgery.
  The concept of the visual analogue scale (VAS), which ranges from minimum score as 0 = no pain and maximum pain score as 10 = worst pain.
  After the herniorrhaphy surgery, the patients will be record pain score by visual analog scale at 4 hours after herniorrhaphy surgery. For patients who have more than 3 point of pain score, parenteral opioid will be perform.

SECONDARY OUTCOMES:
Wound hematoma | 24 hours
  Abnormal bleeding at surgical wound.

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Director — 270, Rama VI road, Ratchathevi, Deapartment of Surgery, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand, 10400; Worasit Chaimongkhalanon, MD, Principal Investigator — 270, Rama VI road, Ratchathevi, Deapartment of Surgery, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand, 10400; Chumpon Wilasrusmee, MD, Principal Investigator — 270, Rama VI road, Ratchathevi, Deapartment of Surgery, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand, 10400
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No